CLINICAL TRIAL: NCT05514210
Title: Feasibility and Effectiveness of a Real-time Heart Team Approach in Complex Coronary Artery Disease
Brief Title: Feasibility and Effectiveness of a Real-time Heart Team Approach in Complex CAD
Acronym: EHEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-1749
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease; Multidisciplinary Communication
Keywords: Complex coronary artery disease; Revascularization decision-making; Heart team process optimization
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real-time heart team group (Experimental): Patients randomized to this group will be accessed and discussed by multidisciplinary specialists during the coronary angiography process
  Interventions: Behavioral: heart team meeting and discussion
- conventional heart team group (Active Comparator): Patients randomized to this group will be accessed and discussed offline and face-to-face by multidisciplinary specialists after the coronary angiography process
  Interventions: Behavioral: heart team meeting and discussion

INTERVENTIONS:
Behavioral: heart team meeting and discussion — When the patient is eligible for the study, the interventional cardiologist will invite a cardiac surgeon to conduct a heart team discussion. Both specialists will assess the patient comprehensively and make an optimal decision for the patient, with consideration patient's preference.

SUMMARY:
This study is aimed to evaluate the clinical outcomes, efficiency and feasibility of the real-time heart team approach and the conventional heart team approach.

DETAILED DESCRIPTION:
This study is a multicenter, randomized controlled trial. According to the inclusion and exclusion criteria, patients with complex coronary artery disease undergoing elective coronary angiography will be prospectively enrolled in the study. Patients will be randomly assigned to the real-time heart team group and the conventional heart team group by block randomization. The real-time heart team group needs to conduct multidisciplinary heart team discussion during the coronary angiography process, while the traditional heart team group needs to conduct multidisciplinary heart team discussion offline and face-to-face after the coronary angiography process. This study will prospectively collect the patient information, heart team meeting process, clinical treatment, and clinical outcomes to evaluate the efficiency and feasibility and differences in clinical outcomes of patients under different heart team approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Significant stenosis in the left main or left main equivalent with or without stenosis in one of the other vessels[Significant stenosis is defined as: 1) a diameter stenosis of at least 50% reduction in luminal diameter by visual assessment or 2) any total occlusion (no age limitation and no exclusion of unfavorable anatomic features); Left main equivalent disease is defined as significant stenosis of the ostium of the left anterior descending and the ostium of the left circumflex.]
2. At least 1 significant stenosis (≥ 70% obstruction) in all 3 major epicardial territories supplying viable myocardium;
3. Other conditions that the interventional cardiologist considers necessary to discuss with cardiac surgeons due to technical and risk considerations.

Exclusion Criteria:

1. Less than 18 years of age;
2. Previous history of PCI or CABG;
3. Admitted for AMI, ECG and biomarker detection indicated acute stage;
4. Patients with severe heart valvular disease, major vascular disease, and giant ventricular aneurysm require surgical treatment;
5. Combined with AF or severe arrhythmia;
6. Other patients admitted to hospital due to emergency circumstances who are not suitable to wait for elective revascularization;
7. Rejection or exclusion of a revascularization mode (PCI or CABG);
8. Refuse to participate in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
1-year major adverse cardiovascular and cerebrovascular events | At 1 year after the coronary angiography
  a composite of all-cause mortality, myocardial infarction, stroke, unplanned revascularization, readmission due to reangina.

SECONDARY OUTCOMES:
time interval between the completion of coronary angiography and the final treatment | through treatment completion, an average of 60 days
  time interval is considered as a key secondary outcome
revascularization decision-making | through study completion, an average of 1 year
  to assess the distribution of the revascularization decision-making made jointly by the heart team and the patients, such as CABG, PCI or medical therapy
revascularization decision-making guideline adherence | through study completion, an average of 1 year
  adjudicated according to 2018 European Society of Cardiology (ESC)/ European Association for Cardio-Thoracic Surgery (EACTS) guideline
heart team decision-making | through study completion, an average of 1 year
  to assess the distribution of the decision-making made by the heart team, such as CABG, PCI or medical therapy
workload of heart team specialists | through study completion, an average of 1 year
  to assess the workload of the specialists participating in the heart team meetings by NASA-TLX scale
success rate of heart team organization | through study completion, an average of 1 year
  to assess the successful-connection with cardiac surgeons during or after the coronary angiography
length of stay | through study completion, an average of 1 year
  to assess length of stay (LOS) before the final treatment, and the totol LOS in hospital
total cost | through study completion, an average of 3 year
  to assess the total cost in hospital for the initial hospitalization and rehospitalization
individual clinical adverse events | At 1 year after the coronary angiography
  including all-cause death, cardiac death, myocardial infarction, stroke, revascularization of target vessels or transplanted vessels, revascularization for any reason, be admitted to hospital with angina again, readmission for cardiac reasons and readmission for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Zheng, MD,PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Su X, Ma H, Lin S, Dou K, Zheng Z. Safety and feasibility of a real-time electronic heart team decision-making approach in patients with complex coronary artery disease: a protocol for a randomised controlled trial (EHEART trial). BMJ Open. 2023 Nov 21;13(11):e076864. doi: 10.1136/bmjopen-2023-076864. PMID 37989362